CLINICAL TRIAL: NCT00709865
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Safety and Tolerability of Intravenous Tonapofylline in Subjects With Acute Decompensated Heart Failure and Renal Insufficiency
Brief Title: Study to Assess the Safety and Tolerability of IV Tonapofylline in Subjects With Acute Decompensated Heart Failure (ADHF) and Renal Insufficiency
Acronym: TRIDENT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160HF301
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Renal Insufficiency; Congestive Heart Failure
Keywords: renal insufficiency; diuretic; congestive heart failure; acute decompensated heart failure
MeSH Terms: conditions — Renal Insufficiency; Heart Failure | interventions — BG 9928; 1,3-dipropyl-8-(2-(5,6-epoxy)norbornyl)xanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): .03 mg/kg
  Interventions: Drug: tonapofylline
- 2 (Experimental): .15 mg/kg
  Interventions: Drug: tonapofylline
- 3 (Experimental): .3 mg/kg
  Interventions: Drug: tonapofylline
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tonapofylline — IV
  Other Names: Adentri; BG9928
  Arms: 1; 2; 3
Drug: Placebo — IV
  Arms: 4

SUMMARY:
The purpose of the current study is to assess the safety and tolerability of intravenous tonapofylline.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of heart failure.
* Must have ADHF, requiring hospitalization, with clinical evidence for volume overload

Exclusion Criteria:

* History of an allergic reaction to any xanthine-containing substance.
* History of seizure
* History of stroke
* Myocardial infarction
* Uncorrected hemodynamically significant primary valvular disease or known Obstructive or restrictive cardiomyopathy.
* Serious systemic infection
* Major surgical procedures within 30 days
* Acute coronary syndrome
* Cardiogenic shock
* Baseline body weight >150 kg
* Participation in any other investigational study of drugs or devices within 30 days prior to Screening
* Nursing mothers, pregnant women, or women planning on becoming pregnant during the study
* Presence of any clinically significant condition that might interfere with optimal safe participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2008-07-31 (Actual); Primary Completion 2009-10-30 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Assess the safety andtolerability of intravenous tonapofylline, when added to standard therapy in subjects hospitalized with ADHF and renal insufficiency. | 0-60 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (166):
- United States (67):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Fort Smith, Arkansas
  - Beverly Hills, California
  - Chula Vista, California
  - Mission Viejo, California
  - Monterey Park, California
  - Oceanside, California
  - Redondo Beach, California
  - San Diego, California
  - Sylmar, California
  - Torrance, California
  - Yuba City, California
  - Hartford, Connecticut
  - Jacksonville, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Lombard, Illinois
  - Indianapolis, Indiana
  - Muncie, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - Ayer, Massachusetts
  - Boston, Massachusetts
  - Hyannis, Massachusetts
  - Springfield, Massachusetts
  - West Springfield, Massachusetts
  - Traverse City, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Lee's Summit, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Ridgewood, New Jersey
  - Johnson City, New York
  - Mineola, New York
  - New York, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Concord, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Camp Hill, Pennsylvania
  - Danville, Pennsylvania
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Orangeburg, South Carolina
  - Nashville, Tennessee
  - Oak Ridge, Tennessee
  - Tullahoma, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Whitney, Texas
  - Danville, Virginia
  - Olympia, Washington
  - Tacoma, Washington
  - Charleston, West Virginia
- Argentina (9):
  - Buenos Aires, BUE
  - Capital Federal, CBA
  - Corrientes, COR
  - Córdoba, CRD
  - Villa Cabrera, CRD
  - Santa Fe, SFE
  - San Luis, SLS
  - San Miguel de Tucumán, TUC
  - Capital Federal
- Australia (5):
  - Darlinghurst, New South Wales
  - Liverpool, New South Wales
  - Canberra
  - Dandenong
  - Melbourne
- Brazil (9):
  - Fortaleza, Ceará
  - Porto Alegre, Rio Grande do Sul
  - Aracaju, Sergipe
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
  - Campo Grande
  - Curitiba
  - Porto Alegre
  - Recife
- Bulgaria (3):
  - Pazardzhik
  - Pleven
  - Sofia
- Canada (2):
  - Vancouver, British Columbia
  - Saint John, New Brunswick
- Czechia (2):
  - Kolín
  - Uherské Hradiště
- Finland (5):
  - Hus
  - Lahti
  - Oulu
  - Seinäjoki
  - Turku
- France (10):
  - Albi
  - Antony
  - Caen
  - Cholet
  - Paris
  - Poitiers
  - Pontoise
  - Strasbourg
  - Toulouse
  - Tourcoinq
- Germany (10):
  - Frankfurt am Main, Hesse
  - Bad Nauheim
  - Berlin
  - Bochum
  - Essen
  - Frankfurt
  - Göttingen
  - Leipzig
  - Regensburg
  - Wuppertal
- India (9):
  - Bangalore, Karna
  - Pune, Mahara
  - New Delhi, National Capital Territory of Delhi
  - Bangalore
  - Bikaner
  - Chennai
  - Delhi
  - Indore
  - Thrissur
- Israel (11):
  - Ashkelon
  - Beer Yaakov
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Petah Tikva
  - Safed
  - Tel Aviv
- Italy (3):
  - Mantova
  - Milan
  - Pavia
- Netherlands (3):
  - Maastricht
  - The Hague
  - Zwolle
- Poland (6):
  - Kościerzyna
  - Olsztyn
  - Słupsk
  - Tarnów
  - Warsaw
  - Wroclaw
- Romania (2):
  - Bacau
  - Bucharest
- Russia (8):
  - Barnaul
  - Kemerovo
  - Krasnoyarsk
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Saratov
  - Tomsk
- Sweden (2):
  - Gothenburg
  - Lidköping